CLINICAL TRIAL: NCT01252043
Title: Retrospective Review of Computed Tomography and Magnetic Resonance Images in Pediatric Patients With Cholestasis
Brief Title: Retrospective Review of CT and MR in Pediatric Patients With Cholestasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Steven Shinn-Forng Peng, staff of Department of Medical Imaging, National Taiwan University Hospital
Other Study IDs: 201010044R
Record Dates: First submitted 2010-11-25; First posted 2010-12-02 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-11

CONDITIONS: Cholestasis; Children
Keywords: cholestasis; children
MeSH Terms: conditions — Cholestasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- cohort: cholestatic children without esophageal variceal bleeding
- study: cholestatic children with esophageal variceal bleeding
- cholestatic children without EV: cholestatic children without esophageal variceal bleeding

SUMMARY:
The investigators will try to predict the risk of esophageal varices (EVs) in long-term BA survivors using noninvasive computed tomography (CT) or magnetic resonance (MR) indices and the measurement of transverse diameters of paraesophageal and gastroesophageal veins.

DETAILED DESCRIPTION:
We intend to review retrospectively 80 pediatric patients on an average of 2 years, who underwent 64-slice CT or MR examinations between January 2005 and Oct 2010 and had EVs on esophagogastroduodenoscopy. Splenic diameters (mm) and hepatic diameters of all patients were measured. Splenic and hepatic volume indices also calculated. The transverse diameters of paraesophageal varices (PVs) and perigastric varices (PGVs) were measured adjacent to the lower thoracic esophagus and within the lesser sac, respectively.

We will try to find out the possible splenic, hepatic or vascular predicting factors useful to evaluate the risk of clinically evident esophageal varices.

ELIGIBILITY:
Inclusion Criteria:

* all cholestatic children with CT, MR and complete medical record

Exclusion Criteria:

* all cholestatic children without either CT, MR or complete medical record

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: younger than 18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
esophageal variceal bleeding | retrospective review

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany TF Shih, M.D., Study Chair — Department of Medical Imaging, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan